CLINICAL TRIAL: NCT01009411
Title: Physiological Study of the Active Stage of Labor
Brief Title: Labor Progress Indices and the Dynamics of the Individual Contraction During the Active Stage of Labor
Status: Completed | Type: Observational
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Collaborators: Barnev Ltd (Other)
Responsible Party: Principal Investigator, Prof. Jacob Bornstein, Chairman, Obstetrics and Gynecology, Western Galilee Hospital-Nahariya
Other Study IDs: BT-1-IS-001
Record Dates: First submitted 2009-10-20; First posted 2009-11-06 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Labor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Control: Patients in active phase of labor not augmented
- Augmented: Augmentation leading to normal progress
- Caesarean section: Augmentation leading to Caesarean section

SUMMARY:
Objective of the study: to obtain new data on the dynamics of the labor process, cervix dilatation and head station on the labor process and to develop a new progress indices.

Background: the best method used today to supervise the labor process is to follow cervix dilatation and head station. Today, the physician or the midwife use manual examination to estimate cervix dilatation and head station. This examination is perform many times in a normal labor process, and even more if there is any delay. The information from these examinations is inaccurate and non-continuous. In case of delay in the labor process, the delay will diagnosed late, because the frequency of the manual examination is about once an hour.

With the assistance of the BirthTrack device we can get continuous data on the labor process and get indices to estimate the labor process progress without the use of vaginal (manual) examination.

40 women in an active labor will take part in the study.

Method: by connecting sensors to the woman abdomen, to the cervix and to the baby head we follow the cervix dilatation and the fetus head station.

ELIGIBILITY:
Inclusion Criteria:

1. Nulliparous women 18 years or older admitted to the labor and delivery unit in active labor (3cm dilatation and contractions).
2. Parturients with epidural anesthesia
3. Singleton fetus in vertex presentation
4. Gestational age 37 or more
5. Reassuring fetal heart tracing
6. The woman is able to read and understand the consent form

Exclusion Criteria:

1. Parturients in natural birth without epidural anesthesia
2. Low lying placenta
3. Known or suspected fetal or maternal infection
4. Maternal thrombocytopenia
5. Maternal bleeding disorder
6. Known major fetal malformation
7. Suspected fetal growth restriction
8. Subjects with significant psychiatric history
9. Subjects with indication for immediate delivery
10. Maternal History of HIV and/or blood transmitted hepatitis and/or active genital Herpes

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Nulliparous women over 18 years admitted to the labor in active labor
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2010-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Birth Track measurements versus manual measurements | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Ofer Barnea, Phd., Study Chair — Barnev Ltd; Prof. Ofer Barnea, Phd., Study Director — Barnev Ltd
Locations (1):
- Westren Gallilie Hospital, Nahariya, Israel